CLINICAL TRIAL: NCT04807179
Title: Prospective Clinical Study To Evaluate The Efficacy And Safety Of An Alexandrite Laser Device For The Treatment Of Acne Scars
Brief Title: Clinical Study to Evaluate Alexandrite Laser for the Treatment of Acne Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7012-RGPL-2021
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Acne Scars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Alexandrite Laser (Experimental): Single arm, self-controlled
  Interventions: Device: Experimental: RF Device Arm

INTERVENTIONS:
Device: Experimental: RF Device Arm — Non-invasive radiofrequency Alexandrite laser

SUMMARY:
The intended use of the Alexandrite laser device used in this study is to assess the efficacy and safety of the Alexandrite laser device for the treatment of acne scars on skin types V and VI.

DETAILED DESCRIPTION:
Subjects are to be enrolled in this clinical study if they are 18-65 years old. A maximum of 25 subjects will be enrolled at 1 study center. Subjects will receive up to 6 treatments (minimum of 4 treatment visits with an optional 5th and 6th treatment) on the face. Subjects will return for follow up visits at 30 and 90 days post last treatment. All subjects will receive a phone call 1 week after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 - 65 years of age.
* Has acne scars on the face (left, right, or front) and willing to undergo treatments with the study device.
* Is a skin type V or VI.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is hypersensitive to light in the near infrared wavelength region.
* The subject takes medication which is known to increase sensitivity to sunlight.
* The subject has seizure disorders triggered by light.
* The subject takes or has taken oral isotretinoin, such as Accutane®, within the last six months.
* The subject has an active localized or systemic infection, or an open wound in area being treated.
* The subject has a significant systemic illness, such as lupus, or an illness localized in area being treated.
* The subject has common acquired nevi that are predisposed to the development of malignant melanoma.
* The subject has herpes simplex in the area being treated.
* The subject is receiving or has received gold therapy.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months to entering this study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Cautionary Criteria:

* The subject has had unprotected sun exposure within four weeks of treatment, including the use of tanning beds or tanning products, such as creams, lotions and sprays.
* The subject has a history of immunosuppression/immune deficiency or an auto-immune disorder.
* The subject has a coagulation disorder or currently using anticoagulation medication, including heavy use of aspirin.
* The subject is taking medications that alter the wound-healing response or evidence of compromised wound healing.
* The subject is known to have a history of keloid formation.
* The subject has a history of skin cancer or suspicious lesions in the treatment area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
Photographic Evaluation of Changes in Treatment Areas | Baseline and 90 day follow up
  Photographic evaluation with ECCA (échelle d'évaluation clinique des cicatrices d'acné) grading comparing pre-treatment images to the 90 day follow up images performed by independent reviewers. This scale gives higher scores based on the number of scars, with the description of the scars determining the weighting factor. The scale ranges from 0 to 540, with a lower score meaning less severe scarring.

SECONDARY OUTCOMES:
Photographic Evaluation of Treatment Areas | Baseline and 30 day follow up
  Photographic evaluation with ECCA (échelle d'évaluation clinique des cicatrices d'acné) grading comparing pre-treatment images to the 30 day follow up images performed by independent reviewers. This scale gives higher scores based on the number of scars, with the description of the scars determining the weighting factor. The scale ranges from 0 to 540, with a lower score meaning less severe scarring.
Blinded evaluation of pre-treatment images vs. follow up images to determine which image is which | Baseline and 30 day follow up
  Blind identification of pre-treatment images vs. 30 day follow up images performed by independent reviewers.
Blinded evaluation of pre-treatment images vs. follow up images to determine which image is which | Baseline and 90 day follow up
  Blind identification of pre-treatment images vs. 90 day follow up images performed by independent reviewers.
Principle Investigator assessment using the Global Aesthetic Improvement Scale (PGAIS) | Baseline and 30 day follow up
  Principle Investigator assessment using the Global Aesthetic Improvement Scale (PGAIS) at the 30 day follow up visit. The GAIS scale ranges from 1 to 5, with 1 being "very much improved," 2 being "much improved," 3 being "improved," 4 being "no change," and 5 being "worse."
Principle Investigator assessment using the Global Aesthetic Improvement Scale (PGAIS) | Baseline and 90 day follow up
  Principle Investigator assessment using the Global Aesthetic Improvement Scale (PGAIS) at the 90 day follow up visit. The GAIS scale ranges from 1 to 5, with 1 being "very much improved," 2 being "much improved," 3 being "improved," 4 being "no change," and 5 being "worse."
Subject assessment using the Global Aesthetic Improvement Scale (SGAIS) | Baseline and 30 day follow up
  Subject assessment using the Global Aesthetic Improvement Scale (SGAIS) at the 30 follow up visit. The GAIS scale ranges from 1 to 5, with 1 being "very much improved," 2 being "much improved," 3 being "improved," 4 being "no change," and 5 being "worse."
Subject assessment using the Global Aesthetic Improvement Scale (SGAIS) | Baseline and 90 day follow up
  Subject assessment using the Global Aesthetic Improvement Scale (SGAIS) at the 90 follow up visit. The GAIS scale ranges from 1 to 5, with 1 being "very much improved," 2 being "much improved," 3 being "improved," 4 being "no change," and 5 being "worse."
Subject satisfaction | 30 day follow up
  Subject satisfaction rates at the 30 day follow up visit. The subject satisfaction scale ranges from 1 to 6, with 1 being extremely unsatisfied, 2 being dissatisfied, 3 being slightly unsatisfied, 4 being slightly satisfied, 5 being satisfied, and 6 being extremely satisfied.
Subject satisfaction | 90 day follow up
  Subject satisfaction rates at the 90 day follow up visit. The subject satisfaction scale ranges from 1 to 6, with 1 being extremely unsatisfied, 2 being dissatisfied, 3 being slightly unsatisfied, 4 being slightly satisfied, 5 being satisfied, and 6 being extremely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (2):
- United States (2):
  - Wallace Skin and Body Institute, Los Angeles, California
  - Laser & Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No